CLINICAL TRIAL: NCT05399355
Title: Pulsed Electromagnetic Fields for Postoperative Analgesia: A Randomized, Triple-Masked, Sham-Controlled Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEMF Surgical Pilot
Record Dates: First submitted 2022-05-19; First posted 2022-06-01 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: Randomized, Triple-Masked, Placebo-Controlled, Parallel-Arm Human Subjects Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigational Drug Service will create the randomization tables and provide the investigators with the appropriate device (active or sham), leaving all participants, investigators, and the statistician masked to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Pulsed Shortwave Treatment with BioElectronics Model 088 (Active Comparator): Application of 7-30 days of nonthermal, pulsed shortwave (radiofrequency) therapy with BioElectronics Model 088
  Interventions: Device: Active Pulsed Shortwave Treatment with BioElectronics Model 088
- Sham Treatment (Sham Comparator): Application of 7-30 days of a nonfunctional sham device.
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Active Pulsed Shortwave Treatment with BioElectronics Model 088 — Application of 7-30 days of nonthermal, pulsed shortwave (radiofrequency) therapy with BioElectronics Model 088
  Other Names: nonthermal, pulsed shortwave (radiofrequency) therapy; pulsed electromagnetic fields therapy
  Arms: Active Pulsed Shortwave Treatment with BioElectronics Model 088
Device: Sham Treatment — Application of 7-30 days of a nonfunctional sham device(s)
  Other Names: Placebo treatment
  Arms: Sham Treatment

SUMMARY:
Pulsed electromagnetic field therapy is a possible method of pain control involving the application of electromagnetic energy (also termed nonthermal, pulsed, shortwave radiofrequency therapy). Food and Drug Administration-cleared devices have been in clinical use for over 70 years. For decades, available devices consisted of a large signal generator and bulky coil applicator that were not portable and produced significant electromagnetic interference, making them impractical for common use. However, small, lightweight, relatively inexpensive, noninvasive, Food and Drug Administration-cleared devices that function for 30 days are now available to treat acute and chronic pain, decrease inflammation and edema, and hasten wound healing and bone regeneration. Therefore, it has the potential to concurrently improve analgesia and decrease or even negate opioid requirements, only without the limitations of opioids and peripheral nerve blocks. The purpose of this pilot study is to explore the possibility of treating acute postoperative pain with nonthermal, pulsed shortwave (radiofrequency) therapy, optimize the study protocol, and estimate the treatment effect in preparation for developing subsequent definitive clinical trials.

DETAILED DESCRIPTION:
The proposed study will be a randomized, participant- and observer-masked, sham-controlled, parallel-arm, human participants pilot study with two primary aims:

Specific Aim 1: To determine the feasibility and optimize the protocol for subsequent clinical trials that will compare the addition of nonthermal, pulsed shortwave therapy to usual and customary analgesia following moderate-to-severely painful surgical procedures.

Specific Aim 2: To estimate the treatment effect of adding nonthermal, pulsed shortwave therapy to usual and customary analgesia on pain and opioid consumption following moderate-to-severely painful surgical procedures. This will provide an idea of the optimal surgical procedures amenable to this analgesic technique and allow determination of the required sample sizes of subsequent definitive clinical trials.

Hypothesis 1: Nonthermal, pulsed shortwave therapy decreases pain in the 7 days following moderate-to-severely painful surgical procedures.

Hypothesis 2: Nonthermal, pulsed shortwave therapy decreases opioid use in the 7 days following moderate-to-severely painful surgical procedures.

This will be a single-center (University of California San Diego), randomized, participant- and observer-masked, sham-controlled, parallel-arm human subjects pilot study.

Enrollment. Participants will be consenting adults undergoing various surgical procedures usually resulting in moderate-to-severe postoperative pain. Study inclusion will be proposed to eligible presurgical patients. If an individual desires study participation, written, informed consent will be obtained using a current University of California San Diego Institutional Review Board-approved informed consent form. The study population of interest includes adult women and men of all races, ethnicity, sexual identity, and socioeconomic status.

Procedures. Following written, informed consent, we will record baseline anthropometric information (age, sex, height, weight, amputation details and current pain levels). Participants will receive any standard peripheral nerve block(s) administered using bupivacaine or ropivacaine 0.5% with epinephrine (standard at University of California San Diego) prior to undergoing their surgical procedure per standard of care.

Treatment Group Assignment. Each participant will be randomized to one of two treatment groups: Active or Sham treatment. There are sham devices produced that are identical to active devices, only they do not deliver pulsed electromagnetic energy. Randomization will be stratified by surgical procedure in block sizes of 2. The computer-generated randomization lists will be created by the University of California San Diego Investigational Drug Service in a 1:1 treatment group ratio using opaque envelopes. The active and sham devices are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff other than the individual who opens the randomization envelope and chooses a sham or active device will be masked to treatment group assignment for the duration of the data collection period. An Investigational Drug Service pharmacist will open the envelope and provide the investigators with the appropriate device, keeping all investigators masked to treatment group assignment. Upon completion of data collection for a specific subgroup (e.g., amputees, total knee arthroplasty), the pharmacist will provide the investigators with a masked list of the treatment groups (e.g., "Treatment A" and "Treatment B"), and the active/sham lists only following analysis for that subgroup, resulting in a triple-masked study (investigators, participants, statistician).

Study intervention. The pulsed shortwave device (2 devices, if there are multiple incisions or the incision is larger than the device diameter; 3 devices for total knee and hip arthroplasty or spinal surgery) will be affixed over the primary wound area(s) using tape and activated prior to recovery room discharge (Experimental). The optimal location to treat phantom pain is currently unknown and will partially informed by the results of this pilot study, and patients will be encouraged to move the devices to a new anatomic location until relief is optimized.

Supplemental analgesics. In addition to the pulsed shortwave device(s), participants will receive standard-of-care supplemental analgesics which can include acetaminophen, ibuprofen, ketorolac, opioids, gabapentin (this is provider- and patient-dependent). Therefore, all patients of this study-regardless of the treatment arm they are randomized to-will continue to receive current usual and customary analgesia: all will receive the same combination of supplemental analgesics they would regardless of study participation. Participants (and their caretakers) will be provided with verbal and written instructions, and the telephone and pager numbers of an investigator available during business hours throughout the treatment period. Participants can shower with the device in place, but not submerge it during swimming or a bath, as advised by the manufacturer.

Participants will be discharged with their pulsed shortwave device(s) in situ and a prescription for immediate-release oral opioid, preferably oxycodone 5 mg tablets, taken for breakthrough pain (surgeons occasionally prefer a different type of opioids such as hydrocodone, which is why we analyze the data using oral oxycodone equivalents). The pulsed shortwave devices will be removed by participants at home following Day 30 when the battery is exhausted (participants may remove them as early as Day 7, if they desire). Removing the devices encompasses tape removal and discarding in the trash (these are disposable, single-use devices).

Of note, if a device is reported lost or nonfunctional during the study, it will be replaced by the investigators by mail if more than 7 days of treatment remain.

Study outcomes: This is an exploratory pilot study to assist in planning subsequent definitive trials and we therefore have no data analysis plan. We will enroll convenience samples for each of the surgical procedures of up to 30 participants for each procedure, and anticipate analyzing each surgical procedure separately from the others. The two outcomes of primary interest will be (1) the "average" and "worst" pain measured with the Numeric Rating Scale (included in the Brief Pain Inventory pain domain), and (2) opioid consumption within the first 7 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

Adult patients of at least 18 years of age undergoing one of these primary surgical procedures:

1. non-mastectomy breast surgery with a single-injection paravertebral nerve block
2. laparoscopic cholecystectomy
3. laparoscopic sleeve gastrectomy
4. percutaneous nephrolithotomy
5. ventral hernia repair
6. inguinal hernia repair
7. knee or hip arthroplasty
8. foot/ankle surgery with at least moderate pain anticipated
9. shoulder acromioclavicular joint repair, labral repair, subacromial decompression, or Bankart repair (without rotator cuff repair)
10. hand/forearm/elbow surgery with at least moderate pain anticipated
11. spinal surgery with at least moderate pain anticipated

Exclusion Criteria:

* concurrent use of an implanted pulse generator (e.g., cardiac pacemaker)
* pregnancy
* incarceration
* chronic opioid/tramadol use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* neuro-muscular deficit of the surgical area/limb
* a planned postoperative perineural local anesthetic infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
per reasonable request and requiring a data sharing agreement
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication of the final dataset.
Access Criteria: contact the Principal Investigator, Dr. Brian Ilfeld

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Started | 59 | 60
Completed | 59 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (15) | 59 (16) | 58 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 44 | 78
  Male | 25 | 16 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 59 | 60 | 119
Height [Mean (Standard Deviation); unit: cm] | 170 (10) | 169 (10) | 169 (10)
Weight [Mean (Standard Deviation); unit: kg] | 78 (19) | 79 (17) | 78 (18)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27 (5) | 27 (5) | 27 (5)
Surgery duration [Mean (Standard Deviation); unit: minutes] | 86 (29) | 93 (39) | 89 (34)
Breast Surgery [Count of Participants; unit: Participants] | 14 | 15 | 29
Cholecystectomy [Count of Participants; unit: Participants] | 7 | 6 | 13
Hernia [Count of Participants; unit: Participants] | 8 | 9 | 17
Hip arthroplasty [Count of Participants; unit: Participants] | 15 | 15 | 30
Knee arthroplasty [Count of Participants; unit: Participants] | 15 | 15 | 30
Adductor Canal block [Count of Participants; unit: Participants] | 15 | 15 | 30
Paravertebral block [Count of Participants; unit: Participants] | 14 | 15 | 29
Erector spinal plane block [Count of Participants; unit: Participants] | 0 | 1 | 1
Rectus sheath block [Count of Participants; unit: Participants] | 1 | 1 | 2
Transversus abdominis plane block [Count of Participants; unit: Participants] | 0 | 1 | 1
No peripheral nerve block [Count of Participants; unit: Participants] | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will the mean value of daily average pain scores measured with the Numeric Rating Scale
Time Frame: Mean value of the average daily pain measured on postoperative days 1, 2, 3, and 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 2.4 (1.6) | 2.6 (1.7)

2. Primary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will the mean value of daily worst pain scores measured with the Numeric Rating Scale
Time Frame: Mean value of the worst daily pain measured on postoperative days 1, 2, 3, and 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 4.6 (2.0) | 4.7 (2.1)

3. Primary Outcome: Total OPIOID Consumption From Recovery Room Discharge Until the Data Collection Phone Call on Postoperative Day 7 (Measured in Oral Oxycodone Equivalents)
Description: Total opioid consumption from recovery room discharge until the data collection phone call on postoperative day 7 (measured in oral oxycodone equivalents).
Time Frame: Cumulative opioid consumption queried on postoperative days 1, 2, 3, and 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | 21 (24) | 17 (26)

4. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale.
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 2.5 (1.9) | 2.9 (2.1)

5. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 2.7 (2) | 3.2 (2)

6. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 2.2 (1.9) | 2.7 (2.3)

7. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.8 (2) | 1.8 (2.1)

8. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.3 (1.8) | 1 (1.7)

9. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1 (1.8) | .7 (1.4)

10. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .7 (1.3) | .7 (1.4)

11. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 0 (0) | .1 (.5)

12. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 5.1 (2.1) | 5.6 (2.4)

13. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 5.2 (2.4) | 5.7 (2.6)

14. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 4.3 (2.7) | 4.6 (2.7)

15. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 3.6 (2.6) | 3.3 (2.9)

16. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 2.5 (2.6) | 1.9 (2.2)

17. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.6 (2.4) | 1.4 (2)

18. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.3 (2.1) | 1.2 (1.9)

19. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 180
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .3 (1.1) | .4 (1.1)

20. Secondary Outcome: LEAST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .7 (1.6) | .9 (1.6)

21. Secondary Outcome: LEAST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .6 (1.2) | .4 (1.2)

22. Secondary Outcome: LEAST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .5 (1.2) | .3 (1.1)

23. Secondary Outcome: LEAST Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .3 (.8) | .2 (.8)

24. Secondary Outcome: CURRENT Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.6 (1.9) | 1.4 (2.2)

25. Secondary Outcome: CURRENT Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.1 (1.8) | .8 (1.6)

26. Secondary Outcome: CURRENT Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .7 (1.5) | .5 (1.3)

27. Secondary Outcome: CURRENT Pain Measured With the Numeric Rating Scale
Description: as for outcome 4
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .5 (1) | .4 (1.1)

28. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | 1.3 (1.7) | 1 (1.3)

29. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | 1.4 (1.7) | 1 (1.4)

30. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | 1.1 (1.8) | 1.1 (2.2)

31. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | .5 (.9) | .7 (1.5)

32. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | .4 (.9) | .3 (.9)

33. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | .1 (.4) | .2 (.7)

34. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | .2 (.9) | .1 (.4)

35. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 180
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
mg | 0 (0) | 0 (0)

36. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: The Brief pain Inventory short form interference subscale is an instrument specifically designed to assess pain and its impact on physical and emotional functioning using a scale of 0-70. The subscale is comprised of 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. The 7 responses for the 7 questions are totaled, producing a scale of 0-70, with 0 being preferred and 70 indicating worse functioning.
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 2.7 (3.1) | 1.8 (2.8)

37. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: as for outcome 36
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.7 (2.7) | 1.1 (2.3)

38. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: as for outcome 36
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | 1.1 (2.3) | .6 (1.5)

39. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: as for outcome 36
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
score on a scale | .6 (1.5) | .3 (1.1)

40. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .4 (1) | .4 (.9)

41. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .8 (1.9) | .6 (1.4)

42. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .4 (1) | .3 (.6)

43. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .7 (1.7) | .5 (.9)

44. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .8 (1.7) | .2 (.7)

45. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 21
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .4 (1.2) | .1 (.4)

46. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 28
Measure: Mean (Standard Deviation); unit: events of awakening
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
events of awakening | .5 (1.2) | .2 (.6)

47. Secondary Outcome: Hospitalization Duration Measured in Days
Description: Day relative to the day of surgery that patient was discharged from the hospital (e.g., same day is postoperative day 0, while the day following surgery is postoperative day 1) over the first postoperative week. The surgical service determines when patients are to be discharged using their own criteria which are not defined by the study.
Time Frame: One single measure recorded on or following the day of surgery (whichever day patient is discharged)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Days | .3 (.5) | .3 (.5)

48. Secondary Outcome: Passive Flexion (Knee and Hip Arthroplasty Patients Only)
Description: The number of degrees of passive flexion achieved from a neutral position
Time Frame: One measure take at the two-week postoperative check (approximately postoperative day 14)
Population: This data point was not able to be collected as participants did not return to the surgeon's office for measurement at 14 days as originally anticipated
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Day Stopped Using Intervention
Description: Day relative to the day of surgery that patient stopped using the intervention for (e.g., same day is postoperative day 0, while the day following surgery is postoperative day 1)
Time Frame: One single measure recorded following the day of surgery
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Days | 21.3 (7.8) | 23.4 (7.9)

50. Secondary Outcome: Desire Use of Device in Hypothetical Future Surgery?
Description: Would the patient want to use the device for a hypothetical surgery in the future (yes, no, or undecided)?
Time Frame: queried on postoperative day 28
Population: The question regarding the desirability of device use in a hypothetical future surgery was inadvertently excluded from the case report forms.
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Surgical Start as Recorded Using Military Time Format
Description: The time of the surgical incision as recorded using military time format
Time Frame: Intraoperative (within the operating room)
Population: This variable was miscatagorized as an outcome measure, when it was measured PRIOR to randomization following surgery. Therefore, it is captured and reported in the baseline measurements as surgical duration.
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Surgical Stop as Recorded Using Military Time Format
Description: The time of the final suture insertion as recorded using military time format
Time Frame: Intraoperative (within the operating room)
Population: as for outcome 51
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Surgical Duration
Description: The time from surgical start to surgical stop measured in minutes and hours
Time Frame: Intraoperative (within the operating room)
Population: as for outcome 51
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 6 | 3

55. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 6 | 3

56. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 0 | 0

57. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 0 | 0

58. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 0 | 0

59. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 0 | 0

60. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one of the intervention devices since the last phone contact
Time Frame: Postoperative day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
Number analyzed (Participants) | 59 | 60
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 postoperative days
Arm/Group | Active Pulsed Shortwave Treatment With BioElectronics Model 088 | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT05399355/Prot_SAP_001.pdf